CLINICAL TRIAL: NCT01360892
Title: Prediction of Incidence of Liver Cancer or PorTal Hypertension in Patients With Viral Hepatitis by Use of Real-time Tissue Elastography
Brief Title: Prediction of Incidence of Liver Cancer by Use of Real-time Tissue Elastography
Acronym: PICTURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kindai University (Other)
Responsible Party: Japan Liver Oncology Group Organization:, Department of Gastroenterology and Hepatology, Kinki University Faculty of Medicine
Other Study IDs: JLOG1003
Record Dates: First submitted 2011-05-21; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Hepatitis B; Chronic Hepatitis C
Keywords: Hepatitis B virus; Hepatitis C virus; Chronic hepatitis; Liver chlorosis; Liver stiffness; Liver fibrosis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis C, Chronic; Hepatitis B; Hepatitis C; Hepatitis, Chronic; Liver Cirrhosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-center cohort study in which the Real-time Tissue Elastography® measurements will predict prospectively the incidence of hepatocellular carcinoma, the incidence and severity of gastroesophageal varices ascites and decompensated cirrhosis in hepatitis B or C patients.

DETAILED DESCRIPTION:
The aim of this study is to validate the predictive value of Real-time Tissue Elastography® by comparison with serum marker or FibroScan® in chronic hepatitis B or C patients.

Every year and for three years, we performed Real-time Tissue Elastography®, blood sampling, gastrointestinal endoscopy. If in the hospital they can perform FibroScan®, FobroScan® also be performed.

Subjects were also performed ultrasonography (US), computed sonography (CT) or magnetic resonance imaging (MRI) evry four or six months.

The time between the Real-time Tissue Elastography®, blood sampling, gastrointestinal endoscopy and FiroScan® must not exceed four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and at least 20 years of age
* Chronic hepatitis B or Chronic hepatitis C

Exclusion Criteria:

* Evidence or history of hepatocellular carcinoma
* History of alcohol abuse (alcohol intake > 20g/day)
* Pregnant or lactating patients
* Psychosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic hepatitis B or C will be eligible for the study. Subjects with other infectious viral diseases or chronic liver disease are excluded for study enrollment.
  Real-time Tissue Elastography®, serum maker and gastrointestinal endoscopy are performed. If in the hopsital they can perform FibroScan®, FobroScan® also be performed.
  The time between the Real-time Tissue Elastography®, blood sampling, FiroScan® must not exceed four weeks.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of carcinogenesis of hepatocellular carcinoma | every four or six months
  Cumulative incidence of carcinogenesis of hepatocellular carcinoma defined as the time from registration to diagnosis of hepatoceluler carcinomais

SECONDARY OUTCOMES:
Cancer-free survival | every four or six months
  Cancer-free survival is defined as the time from registration to death due to cencer or any cause
Overall survival | one year
  Overall survival is defined as the time from registration to death due to any cause
The cumulative incidence and severity of gastro-esophageal varices | one year
  It is estimated by gastrointestinal scope for every year
The cumulative incidence and severity of decompensated cirrhosis | one year
  Jaundice, ascites, edema and hepatic encephalopathy etc. is evaluated as decompensated cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, Professor, Study Chair — Kinki University Faculty of Medicine
Locations (1):
- Kinki University Faculty of Medicine, Ōsaka-sayama, Osaka, Japan